CLINICAL TRIAL: NCT06024837
Title: Performance of Spectral CT-scan in Patients With Metastatic Colorectal Cancer: a Prospective Multicentre Study
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN1162022/CHUSTE
Record Dates: First submitted 2023-08-21; First posted 2023-09-06 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Colo-rectal Cancer
Keywords: Colo-rectal cancer; spectral CT scan; liver metastases; peritoneal carcinosis
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Colo-rectal Cancer: Patients with Colo-rectal Cancer will be included.
  Interventions: Other: CT Images

INTERVENTIONS:
Other: CT Images — Analysis of CT images of peritoneal and/or liver metastases from colorectal cancer

SUMMARY:
Spectral CT is a rapidly expanding imaging modality that allows a reduction in iodine dose and irradiation compared to conventional scanning. It uses the difference in attenuation of the material according to the two different energy levels of the incident x-ray beams. The dual-energy scanner has a wide range of clinical applications, particularly in abdominal imaging.

DETAILED DESCRIPTION:
First of all, the virtual creation of mono-energy images between 40 and 140 keV has shown subjective and objective improvement of tumor detection of hypovascular lesions using low energies (40keV). It has been shown to be of interest in vascular and cardiac imaging, and to reduce artefacts in bone imaging. However, its performance in oncology analysis has been little studied. The selection of patients for peritoneal and hepatic carcinosis surgery is fundamental, as surgery allows a prolongation of survival, but are associated with a non-negligible morbi-mortality rate.

Spectral CT provides improved detection of peritoneal carcinosis and liver metastases of colorectal cancer compared to conventional CT acquisition.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed for colorectal cancer with synchronous or metachronous liver metastases and/or peritoneal carcinosis
* Patients with a curative surgical resection plan

Exclusion Criteria:

* Patients with non-metastatic colorectal cancer
* Patients treated with chemotherapy without surgical plans
* Patients with colorectal cancer with extra-hepatic and extra-peritoneal metastases alone (e.g. lung, bone)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with synchronous or metachronous peritoneal and/or liver metastases of colorectal cancer with curative surgical plans.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Comparison of peritoneal lesion mapping between spectral scanning and conventional scanning | Year : 1
  Comparison of peritoneal lesion mapping between spectral scanning (monoenergetic acquisitions, iodine mapping, etc.) and conventional scanning (acquisition obtained during spectral acquisition).
Comparison of hepatic lesion mapping between spectral scanning and conventional scanning | Year : 1
  Comparison of hepatic lesion mapping between spectral scanning (monoenergetic acquisitions, iodine mapping, etc.) and conventional scanning (acquisition obtained during spectral acquisition).

SECONDARY OUTCOMES:
Evaluation of response to chemotherapy in RECIST 1.1 | Year : 1
  Collection of demographic, biological and surgical data.
Evaluation of response to chemotherapy in Radiomics | Year : 1
  Collection of demographic, biological and surgical data.

CONTACTS AND LOCATIONS:
Overall Officials: Rémi GRANGE, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No